CLINICAL TRIAL: NCT00005122
Title: Evans County Studies
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 901; R37HL003341 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2000-06

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Myocardial Infarction; Angina Pectoris; Cerebrovascular Accident; Coronary Disease; Ischemic Attack, Transient
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Myocardial Infarction; Angina Pectoris; Stroke; Coronary Disease; Ischemic Attack, Transient

SUMMARY:
To conduct surveillance of cardiovascular morbidity and mortality and its correlation with known risk factors in all cohort study groups in Evans County, Georgia.

DETAILED DESCRIPTION:
BACKGROUND:

The Evans County Studies were initiated as a result of a request from the National Heart Institute in the late 1950's to develop epidemiological studies in areas where significant racial or ethnic differences in cardiovascular disease rates had been observed and where a stable population was available for long-term follow-up. Evans County was in a region of the United States known, at the time, to have the highest total death rates for all causes, of which coronary heart disease and hypertension were major contributors. At that time, Black males and females were known to have four times less coronary heart disease than white males, showed no sex differences for coronary heart disease mortality, and consumed more animal fat and had 50 percent more hypertension.

In 1960, the original Evans County Study cohort was formed when 92 percent of all residents, Black and white, aged 40-74 years and a 50 percent sample of residents aged 15-39 years were given a complete physical examination and a variety of laboratory tests. The major purpose of the original study was to determine factors associated with coronary and related cardiovascular diseases and to explain the low frequency of coronary heart disease in Blacks. Of the initial cohort of 3,102 individuals in 1960, approximately 2,500 were re-examined from 1967 to 1969. Variables studied included serum lipid levels, blood pressure, blood clotting factors, catecholamine levels, physical activity, and social, psychological, and economic factors. Necropsy data were also collected. Follow-up continued on the remaining cohort of approximately 1,900.

Over the years many additional studies were added. The Lipoprotein Phenotyping Study examined which fraction or fractions of high density lipoproteins or low density lipoproteins were related to increased risk for coronary heart disease. The Black-White Neonatal Blood Pressure Study related blood pressure levels during the first year of life to the subsequent development of hypertension and comparing similar groups in other geographical areas to the Evans County group. The Contraceptive Steroids on Blood Pressure Study, funded by the National Institute of Child Health and Human Development, related antecedent characteristics to the development of hypertension or thrombotic disease in the first time oral contraceptive user. The Evans County Health Department also participated Hypertension Detection and Followup Program clinical trial and continued surveillance of the cohort.

Other studies included: the use of defined biracial pedigree cohorts as genetic models to define the possible inheritance of hypertension, hyperlipidemias, coronary heart disease, and thrombosis; maintenance of a collection of frozen sera and food; evaluating new tests to indicate differences in intravascular coagulation between racial and social class groups as related to physical activity, social mobility, and dietary deficiency; studies of the possible relationship to hypertension of dietary sodium-potassium and calcium and selenium intake.

DESIGN NARRATIVE:

Follow-up of the original Evans County Study cohort was achieved by contacting each member annually by mail, telephone, or personal visit, weekly surveys of all admissions at the Evans Memorial Hospital and Statesboro Hospital; survey of daily obituaries in the local newspapers. In the event of a death, autopsy reports and hospital records were obtained. Twice a year teams of consulting neurologists and cardiologists visited Evans County to examine all suspected surviving cases of stroke, transient ischemic attack, myocardial infarction, and angina pectoris. Home visits were conducted for patients who did not visit the medical facility.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1958-07; Study Completion 1995-08 (Actual)

REFERENCES:
- [Background] Fodor JG, Heyden S, Chockalingam A, Logan AG, Hames CG. The P-wave in the electrocardiogram of hypertensive patients before and after therapy. Can J Cardiol. 1986 Sep-Oct;2(5):264-7. PMID 3768785
- [Background] Curb JD, Borhani NO, Blaszkowski TP, Zimbaldi N, Fotiu S, Williams W. Patient-perceived side effects to antihypertensive drugs. Am J Prev Med. 1985 Jan-Feb;1(1):36-40. PMID 3870892
- [Background] Johnson MA, Dooley SP, Caster WO, Hames CG: The Relationship Between Dietary Calcium and Blood Pressure in the Elderly. J Clin Exp Gerontology, 8: (3 & 4), 161-172, 1986
- [Background] Smith DK, Teague RJ, McAdam PA, Feldman DS, Feldman EB. Selenium status of malnourished hospitalized patients. J Am Coll Nutr. 1986;5(3):243-52. doi: 10.1080/07315724.1986.10720128. PMID 3090129
- [Background] Chen XS, Xue A, Morris VC, Ferrans VJ, Herman EH, el-Hage A, Levander OA. Effect of selenium deficiency on the chronic toxicity of adriamycin in rats. J Nutr. 1986 Dec;116(12):2453-65. doi: 10.1093/jn/116.12.2453. PMID 3806242
- [Background] Singh VK, Fudenberg HH. Immunopharmacological approach to the study of chronic brain disorders. Prog Drug Res. 1986;30:345-63. doi: 10.1007/978-3-0348-9311-4_10. No abstract available. PMID 3544047
- [Background] Marazita ML, Elston RC, Namboodiri KK, Hames CG. Genetic analysis of serum lipid levels and blood pressure in a large kindred. Am J Med Genet. 1987 Mar;26(3):511-9. doi: 10.1002/ajmg.1320260302. PMID 3565465
- [Background] Strogatz DS, Tyroler HA, Watkins LO, Hames CG. Electrocardiographic abnormalities and mortality among middle-aged black men and white men of Evans County, Georgia. J Chronic Dis. 1987;40(2):149-55. doi: 10.1016/0021-9681(87)90066-x. PMID 3818868
- [Background] Combs GF, Spallholz JE, Levander OA, Oldfield JE: Selenium in Biology and Medicine, Third lnternational Symposium, Beijing, China. Two Books, Parts A and B, published in 1987
- [Background] Hames CG: An Urgent Methodological Need for Antioxidant Research as Seen by an Epidemiologist. Book, Selenium in Biology and Medicine, 3rd lnterntl Symposium, Beijing, China, Part B, 1987
- [Background] Comberg HU, Knowles M, Tyroler HA, Heyden S, Hames CG, Sabo D. Status of patients seven years after completion of the hypertension detection and follow-up program in Evans County, Georgia. J Natl Med Assoc. 1988 Dec;80(12):1285-92. PMID 3249331
- [Background] Daniels SR, Heiss G, Davis CE, Hames CG, Tyroler HA. Race and sex differences in the correlates of blood pressure change. Hypertension. 1988 Mar;11(3):249-55. doi: 10.1161/01.hyp.11.3.249. PMID 3350588
- [Background] Somervell PD, Kaplan BH, Heiss G, Tyroler HA, Kleinbaum DG, Obrist PA. Psychologic distress as a predictor of mortality. Am J Epidemiol. 1989 Nov;130(5):1013-23. doi: 10.1093/oxfordjournals.aje.a115402. PMID 2816889
- [Background] Humble C, Croft J, Gerber A, Casper M, Hames CG, Tyroler HA. Passive smoking and 20-year cardiovascular disease mortality among nonsmoking wives, Evans County, Georgia. Am J Public Health. 1990 May;80(5):599-601. doi: 10.2105/ajph.80.5.599. PMID 2327539
- [Background] Moorman PG, Hames CG, Tyroler HA. Socioeconomic status and morbidity and mortality in hypertensive blacks. Cardiovasc Clin. 1991;21(3):179-94. PMID 1828391
- [Background] Knapp RG, Keil JE, Sutherland SE, Rust PF, Hames C, Tyroler HA. Skin color and cancer mortality among black men in the Charleston Heart Study. Clin Genet. 1995 Apr;47(4):200-6. doi: 10.1111/j.1399-0004.1995.tb03959.x. PMID 7628122
- [Background] PARKER WC, BEARN AG. Haptoglobin and transferrin variation in humans and primates: two new transferrins in Chinese and Japanese populations. Ann Hum Genet. 1961 Dec;25:227-41. doi: 10.1111/j.1469-1809.1962.tb01523.x. No abstract available. PMID 14483937
- [Background] HAMES CG, GREENBERG BG. A comparative study of serum cholesterol levels in school children and their possible relation to atherogenesis. Am J Public Health Nations Health. 1961 Mar;51(3):374-85. doi: 10.2105/ajph.51.3.374. No abstract available. PMID 13711000
- [Background] WORKMAN PL, BLUMBERG BS, COOPER AJ. SELECTION, GENE MIGRATION AND POLYMORPHIC STABILITY IN A U. S. WHITE AND NEGRO POPULATION. Am J Hum Genet. 1963 Dec;15(4):429-37. No abstract available. PMID 14097237
- [Background] MCDONOUGH JR, HAMES CG, STULB SC, GARRISON GE. CARDIOVASCULAR DISEASE FIELD STUDY IN EVANS COUNTY, GA. Public Health Rep (1896). 1963 Dec;78(12):1051-9. No abstract available. PMID 14090074
- [Background] McDonough JR, Hames CG, Griffin LH, Edwards AJ: Observations on Serum Cholesterol Levels in the Twin Population of Evans County, Ga. Circulation, XXV: June 1963
- [Background] ROBINSON JC, BLUMBERG BS, PIERCE JE, COOPER AJ, HAMES CG. STUDIES ON INHERITED VARIANTS OF BLOOD PROTEINS. II. FAMILIAL SEGREGATION OF TRANSFERRIN B1-2B2. J Lab Clin Med. 1963 Nov;62:762-5. No abstract available. PMID 14078012
- [Background] COOPER AJ, BLUMBERG BS, WORKMAN PL, MCDONOUGH JR. BIOCHEMICAL POLYMORPHIC TRAITS IN A U. S. WHITE AND NEGRO POPULATION. Am J Hum Genet. 1963 Dec;15(4):420-8. No abstract available. PMID 14097236
- [Background] BLUMBERG BS, WORKMAN PL, HIRSCHFELD J. GAMMA-GLOBULIN, GROUP SPECIFIC, AND LIPOPROTEIN GROUPS IN A U.S. WHITE AND NEGRO POPULATION. Nature. 1964 May 9;202:561-3. doi: 10.1038/202561a0. No abstract available. PMID 14195051
- [Background] HAMES CG, MCDONOUGH JR, ELLIOTT JL. HYPERTENSION IN IDENTICAL TWINS. Lancet. 1964 Sep 12;2(7359):585. doi: 10.1016/s0140-6736(64)90648-8. No abstract available. PMID 14172370
- [Background] MCDONOUGH JR, GARRISON GE, HAMES CG. BLOOD PRESSURE AND HYPERTENSIVE DISEASE AMONG NEGROES AND WHITES; A STUDY IN EVANS COUNTY, GEORGIA. Ann Intern Med. 1964 Aug;61:208-28. doi: 10.7326/0003-4819-61-2-208. No abstract available. PMID 14204858
- [Background] KUEPPERS F, BRISCOE WA, BEARN AG. HEREDITARY DEFICIENCY OF SERUM ALPHA-L-ANTITRYPSIN. Science. 1964 Dec 25;146(3652):1678-9. doi: 10.1126/science.146.3652.1678. PMID 14224514
- [Background] Stulb SC, Mcdonough JR, Greenberg BG, Hames CG. THE RELATIONSHIP OF NUTRIENT INTAKE AND EXERCISE TO SERUM CHOLESTEROL LEVELS IN WHITE MALES IN EVANS COUNTY, GEORGIA. Am J Clin Nutr. 1965 Feb;16(6):238-42. doi: 10.1093/ajcn/16.2.238. No abstract available. PMID 14253896
- [Background] MCDONOGH JR, HAMES CG, STULB SC, GARRISON GE. CORONARY HEART DISEASE AMONG NEGROES AND WHITES IN EVANS COUNTY, GEORGIA. J Chronic Dis. 1965 May;18:443-68. No abstract available. PMID 14292191
- [Background] MCDONOUGH JR, HAMES CG, GARRISON GE, STULB SC, LICHTMAN MA, HEFELFINGER DC. THE RELATIONSHIP OF HEMATOCRIT TO CARDIOVASCULAR STATES OF HEALTH IN THE NEGRO AND WHITE POPULATION OF EVANS COUNTY, GEORGIA. J Chronic Dis. 1965 Mar;18:243-57. doi: 10.1016/0021-9681(65)90151-7. No abstract available. PMID 14278160
- [Background] Lichtman MA, Hames CG, Mcdonough JR. SERUM PROTEIN ELECTROPHORETIC FRACTIONS AMONG NEGRO AND WHITE SUBJECT IN EVANS COUNTY, GEORGIA. Am J Clin Nutr. 1965 Jun;16:492-508. doi: 10.1093/ajcn/16.6.492. No abstract available. PMID 14297282
- [Background] Lichtman MA, Hames CG, McDonough JR: Serum Gamma Globulin Levels Among Negroes and Whites in Evans County, Ga. Clin Res, 13:30, 1965
- [Background] Ibrahim MA, Jenkins CD, Cassel JC, McDonough JR, Hames CG. Personality traits and coronary heart disease. Utilization of a cross-sectional study design to test whether a selected psychological profile precedes or follows manifest coronary heart disease. J Chronic Dis. 1966 Mar;19(3):255-71. doi: 10.1016/0021-9681(66)90131-7. No abstract available. PMID 5910969
- [Background] Garrison GE, McDonough JR, Hames CG, Stulb SC. Prevalence of chronic congestive heart failure in the population of Evans County, Georgia. Am J Epidemiol. 1966 Mar;83(2):338-44. doi: 10.1093/oxfordjournals.aje.a120589. No abstract available. PMID 5930780
- [Background] Berg K, Bearn AG. An inherited X-linked serum system in man; the Xm system. J Exp Med. 1966 Feb 1;123(2):379-97. doi: 10.1084/jem.123.2.379. PMID 4159523
- [Background] Skinner JS, Benson H, McDonough JR, Hames CG. Social status, physical activity, and coronary proneness. J Chronic Dis. 1966 Jul;19(7):773-83. doi: 10.1016/0021-9681(66)90075-0. No abstract available. PMID 5965353
- [Background] Hames CG, McDonough JR, Stulb SC, Garrison G: Physical Activity and Ischemic Heart Disease Among Negroes and Whites in Evans County, Ga. Prevention of Ischemic Heart Disease: Principles and Practice by Wilhelm Raab, Charles Thomas, Publisher, 1966
- [Background] Hames CG. Physical activity and coronary heart disease. J Med Assoc Ga. 1967 Jul;56(7):308. No abstract available. PMID 6043924
- [Background] McDonough JR, Hames CG. Influence of race, sex and occupation on seasonal changes in serum cholesterol. Am J Epidemiol. 1967 May;85(3):356-64. doi: 10.1093/oxfordjournals.aje.a120697. No abstract available. PMID 6025080
- [Background] Brewer GJ, Gall JC, Honeyman M, Gershowitz H, Shreffler DC, Dern RJ, Hames C. Inheritance of quantitative expression of erythrocyte glucose-6-phosphate dehydrogenase activity in the negro--a twin study. Biochem Genet. 1967 Jun;1(1):41-53. doi: 10.1007/BF00487735. No abstract available. PMID 5629307
- [Background] Lichtman MA, Vaughan JH, Hames CG. The distribution of serum immunoglobulins, anti-gamma-G globulins ("rheumatoid factors") and antinuclear antibodies in White and Negro subjects in Evans County, Georgia. Arthritis Rheum. 1967 Jun;10(3):204-15. doi: 10.1002/art.1780100306. No abstract available. PMID 4165682
- [Background] McDonough JR, Garrison GE, Hames CG: Blood Pressure and Hypertensive Disease Among Negroes and Whites in Evans County, Ga. In Epidemiology of Hypertension, Grune & Stratton, Inc., 1967
- [Background] Lichtman MA, McDonough JR, Hames CG: Serum Gamma Globulin Concentration in Related and Non-Related Subjects. Hum Biol, 39:No 3, Sept. 1967
- [Background] Kueppers F, Bearn AG. An inherited alpha-1-antitrypsin variant. Humangenetik. 1967 Sep 6;4(3):217-20. doi: 10.1007/BF00292195. No abstract available. PMID 6080804
- [Background] Jenkins CD, Hames CG, Zyzanski SJ, Rosenman RH, Friedman M. Psychological traits and serum lipids. I. Findings from the California Psychological Inventory. Psychosom Med. 1969 Mar-Apr;31(2):115-28. doi: 10.1097/00006842-196903000-00004. No abstract available. PMID 5783999
- [Background] Heyden S, Bartel AG, Hames CG, McDonough JR. Elevated blood pressure levels in adolescents, Evans County, Georgia. Seven-year follow-up of 30 patients and 30 controls. JAMA. 1969 Sep 15;209(11):1683-9. No abstract available. PMID 5394361
- [Background] Hames CG. Coronary heart disease and smoking. A reducible risk factor. J Med Assoc Ga. 1969 Oct;58(10):440. No abstract available. PMID 5346934
- [Background] Hames CG: Inter-Disciplinary Findings of the Evans County Epidemiological Research Project, Workshop-Conference, Fundamental Data on Reactions of Vascular Tissue in Man, Lindau, W. Germany, April 19-25, 1970
- [Background] Bartel AG, Hames CG. Intensive coronary care in a 42-bed rural hospital. J Med Assoc Ga. 1970 Jul;59(7):285-9. No abstract available. PMID 5448263
- [Background] Hames CG: The Correlation of Ischemic Heart Disease with Social Class Among Whites and Blacks in a Total Community Epidemiological Study. Lex et Scientia, 7: No 2, April-June 1970
- [Background] Hames CG. Stress and heart disease. J Med Assoc Ga. 1970 May;59(5):194-5. No abstract available. PMID 5431711
- [Background] Deasy LC. Some reflections on coronary heart disease: socio-medical implications for patients and their families. Soc Sci Med (1967). 1970 Apr;3(4):659-67. doi: 10.1016/0037-7856(70)90033-8. No abstract available. PMID 5478779
- [Background] Heyman A, Karp HR, Heyden S, Bartel A, Cassel JC, Tyroler HA, Hames CG. Cerebrovascular disease in the biracial population of Evans County, Georgia. Arch Intern Med. 1971 Dec;128(6):949-55. No abstract available. PMID 5132454
- [Background] Cassel J, Heyden S, Bartel AG, Kaplan BH, Tyroler HA, Cornoni JC, Hames CG. Occupation and physical activity and coronary heart disease. Arch Intern Med. 1971 Dec;128(6):920-8. No abstract available. PMID 5132450
- [Background] Cassel J, Heyen S, Bartel AG, Kaplan BH, Tyroler HA, Cornoni JC, Hames CG. Incidence of coronary heart disease by ethnic group, social class, and sex. Arch Intern Med. 1971 Dec;128(6):901-6. No abstract available. PMID 5132447
- [Background] Blumberg BS, Hesser JE. Loci differentially affected by selection in two American black populations. Proc Natl Acad Sci U S A. 1971 Oct;68(10):2554-8. doi: 10.1073/pnas.68.10.2554. PMID 5289889
- [Background] Simpson MT, Hames CG, Olewine DA, Ramsey FH, Meier R. Physical activity, catecholamines, and platelet stickiness. Recent Adv Stud Cardiac Struct Metab. 1972;1:742-52. No abstract available. PMID 4681499
- [Background] Farrar WE Jr, Gibbins SD, Whitfield ST. Low prevalence of antibody to Trypanosoma cruzi in Georgia. Am J Trop Med Hyg. 1972 Jul;21(4):404-6. doi: 10.4269/ajtmh.1972.21.404. No abstract available. PMID 4626153
- [Background] Heyden S. [Epidemiology of cerebral vascular occlusions]. Verh Dtsch Ges Inn Med. 1972;78:393-408. No abstract available. German. PMID 4665675
- [Background] Heyden S, Bartel A, Cassel JC, Hames CG, Tyroler HA, Meier R: Physiologische, Pharmakologische Und Klinische Wirkungen Des Kaffees. Supplementum 14, Darmstadt, 1972
- [Background] Karp HR, Heyman A, Heyden S, Bartel AG, Tyroler HA, Hames CG. Transient cerebral ischemia. Prevalence and prognosis in a biracial rural community. JAMA. 1973 Jul 9;225(2):125-8. doi: 10.1001/jama.225.2.125. No abstract available. PMID 4740273
- [Background] Klein R, Klein BE, Cornoni JC, Maready J, Cassel JC, Tyroler HA. Serum uric acid. Its relationship to coronary heart disease risk factors and cardiovascular disease, Evans County, Georgia. Arch Intern Med. 1973 Sep;132(3):401-10. doi: 10.1001/archinte.132.3.401. No abstract available. PMID 4783021
- [Background] Hyden S, Tyroler HA, Hames CG, Bartel A, Thompson JW, Krishan I, Rosenthal T. Diet treatment of obese hypertensives. Clin Sci Mol Med Suppl. 1973 Aug;45 Suppl 1:209s-12. doi: 10.1042/cs045209s. No abstract available. PMID 4593567
- [Background] Hames CG. Hypertension in general practice. Prev Med. 1974 Sep;3(3):313-22. doi: 10.1016/0091-7435(74)90042-5. No abstract available. PMID 4278130
- [Background] Tyroler HA, Heyden S, Hames CG: Weight and Hypertension: Evans County Studies in Blacks and Whites. In Paul O (Ed) Epidemiology and Control of Hypertension, Second International Symposium on the Epidemiology of Hypertension, Chicago Heart Association, 1974
- [Background] Simpson MT, Olewine DA, Jenkins CD, Ramsey FH, Zyzanski SJ, Thomas G, Hames CG. Exercise-induced catecholamines and platelet aggregation in the coronary-prone behavior pattern. Psychosom Med. 1974 Nov-Dec;36(6):476-87. doi: 10.1097/00006842-197411000-00003. No abstract available. PMID 4431856
- [Background] Garrison GE, Gullen WH, Connell CM. Migration of urbanites to small towns for medical care. JAMA. 1974 Feb 18;227(7):770-3. No abstract available. PMID 4405843
- [Background] Hames CG: Most likely to Succeed as a Candidate for a Coronary Attack. New Horizons in Cardiovascular Practice, University Park Press, 1975
- [Background] Heyden S, Hames CG. [Diet therapy of elevated blood pressure values in overweight persons. Hypertension-intervention study: 1 year's report from the Evans-County (Ga.) study]. Med Welt. 1974 Dec 6;25(49):2041-3. No abstract available. German. PMID 4444500
- [Background] Goldberg S, Krishan I, Hames CB, Knight M, Spierto FW. Elevated renin levels in normotensive adolescents. Pediatrics. 1974 Nov;54(5):596-8. No abstract available. PMID 4453457
- [Background] Hames CG. Natural history of essential hypertension in Evans County, Georgia. Postgrad Med. 1974 Nov;56(6):119-25. doi: 10.1080/00325481.1974.11713908. No abstract available. PMID 4427855
- [Background] Johnson AL, Cornoni JC, Cassel JC, Tyroler HA, Heyden S, Hames CG. Influence of race, sex and weight on blood pressure behavior in young adults. Am J Cardiol. 1975 Apr;35(4):523-30. doi: 10.1016/0002-9149(75)90835-8. PMID 1119403
- [Background] Klein B, Klein R, Haseman J, Maready J, Hames C. Corneal arcus and cardiovascular disease in Evans County, Georgia. Arch Intern Med. 1975 Apr;135(4):509-11. PMID 1138662
- [Background] Deubner DC, Tyroler HA, Cassel JC, Hames CG, Becker C. Attributable risk, population attributable risk, and population attributable fraction of death associated with hypertension in a biracial population. Circulation. 1975 Nov;52(5):901-8. doi: 10.1161/01.cir.52.5.901. PMID 1175273
- [Background] Tyroler HA, Hames CG, Krishan I, Heyden S, Cooper G, Cassel JC. Black-white differences in serum lipids and lipoproteins in Evans County. Prev Med. 1975 Dec;4(4):541-9. doi: 10.1016/0091-7435(75)90040-7. No abstract available. PMID 1208366
- [Background] Heyden S: Risk Factors of Ischemic Heart DIsease. Monogram, 1975
- [Background] Gryglewski RJ, Szczeklik A, Bieron K. Morphine antagonises prostaglandin E1- mediated inhibition of human platelet aggregation. Nature. 1975 Jul 3;256(5512):56-7. doi: 10.1038/256056a0. No abstract available. PMID 1134581
- [Background] Jenkins CD, Thomas G, Olewine D, Zyzanski SJ, Simpson MT, Hames CG. Blood platelet aggregation and personality traits. J Human Stress. 1975 Dec;1(4):34-46. doi: 10.1080/0097840X.1975.9939551. PMID 1235120
- [Background] Beaglehole R, Tyroler HA, Cassel JC, Deubner DC, Bartel AG, Hames CG. An epidemiological study of left ventricular hypertrophy in the biracial population of Evans County, Georgia. J Chronic Dis. 1975 Nov;28(10):549-59. doi: 10.1016/0021-9681(75)90061-2. No abstract available. PMID 127804
- [Background] Beaglehole R, Heiss G, Tyroler HA, Cassel JC, Hames CG. Prevalence and incidence data in the assessment of the risk of coronary heart disease. Am J Epidemiol. 1975 Jul;102(1):55-62. doi: 10.1093/oxfordjournals.aje.a112134. PMID 1155437
- [Background] Hames CG: Critique: Diet and Hyperlipidemia as Primary Etiological Factors in Ischemic Heart Disease. Henry I. Russek (Ed) in: Cardiovascular Problems, University Park Press, Baltimore, 1976
- [Background] Hames CG: A Study of Behavioral Modification and Physiological Response Their Possible Relationship to lschemic Heart Disease. Henry I. Russek (Ed) in: Cardiovascular Problems, University Park Press, Baltimore, 1976
- [Background] Berg K, Hames C, Dahlen G, Frick MH, Krishan I. Genetic lipoprotein variation and lipid levels in man. Clin Genet. 1976 Aug;10(2NA-NA-760903-760909):97-103. doi: 10.1111/j.1399-0004.1976.tb00020.x. PMID 954231
- [Background] Berg K, Hames C, Dahlen G, Frick MH, Krishan I. Genetic variation in serum low density lipoproteins and lipid levels in man. Proc Natl Acad Sci U S A. 1976 Mar;73(3):937-40. doi: 10.1073/pnas.73.3.937. PMID 176662
- [Background] Heyden S, Tyroler HA, Cassel JC, Hames CG, Becker C, Heiss G. Coffee consumption and mortality in a community study--Evans Co., Ga. Z Ernahrungswiss. 1976 Jun;15(2):143-50. doi: 10.1007/BF02018434. PMID 969703
- [Background] Olewine DA, Simpson MT, Ramsey FR, Thomas G, Hames CG: Submaximal Exercise Response to Plasma and Urinary Catecholamines in Young Adult Males of Different Aerobic Capacities. Physiologist, 19:(No. 3), August, 1976
- [Background] Chah CC, Caster WO, Combs GF, Hames CG, and Heyden S: Macro and Micro Elements and the Epidemiology of Cardiovascular Disease. Trace Sub in Environ Health X, 1976
- [Background] Greene SB, Aavedal MJ, Tyroler HA, Davis CE, Hames CG. Smoking habits and blood pressure change: a seven year follow-up. J Chronic Dis. 1977 Jul;30(7):401-13. doi: 10.1016/0021-9681(77)90034-0. No abstract available. PMID 885983
- [Background] Castelli WP, Doyle JT, Gordon T, Hames CG, Hjortland MC, Hulley SB, Kagan A, Zukel WJ. HDL cholesterol and other lipids in coronary heart disease. The cooperative lipoprotein phenotyping study. Circulation. 1977 May;55(5):767-72. doi: 10.1161/01.cir.55.5.767. PMID 191215
- [Background] Castelli WP, Doyle JT, Gordon T, Hames CG, Hjortland MC, Hulley SB, Kagan A, Zukel WJ. Alcohol and blood lipids. The cooperative lipoprotein phenotyping study. Lancet. 1977 Jul 23;2(8030):153-5. doi: 10.1016/s0140-6736(77)90176-3. PMID 69778
- [Background] Farmer PK, Olewine DA, Comer DW, Edwards ME, Coleman TM, Thomas G, Hames CG: Frontalis Muscle Tension and Occipital Alpha Production in Young Males with Coronary Prone (Type A) and Coronary Resistant (Type B) Behavior Patterns: Effects of Exercise. Med and Sci in Sports, 10:51, 1978
- [Background] Hames CG, Heyden S, Prineas R, Heiss G, Comberg HU, Sneiderman CH: The Natural History of Hypertension in Evans County, Ga. ln: Athero- sclerosis: Its Pediatric Aspects, Grune & Stratton, 1978
- [Background] Heyden S, Manegold CH, Hames CG, and Patzschke U: Natriumbeschrankung als therapeutische und praventive maBnahme bei Hypertonie. Aktuelle Ernahrungsmedizin, June, 1978
- [Background] Heyden S, Tyroler HA, Heiss G, Hames CG, Bartel A. Coffee consumption and mortality. Total mortality, stroke mortality, and coronary heart disease mortality. Arch Intern Med. 1978 Oct;138(10):1472-5. PMID 708166
- [Background] Olewine DA, Thomas G, Simpson MT, Hames CG: 24 Hour Urinary Steroid Excretion Pattern in Young Males with Type A and Type B Behavior Patterns. Physiologist, 21:4, Aug, 1978
- [Background] Vergroesen AJ, Fleischman AI, Comberg HU, Heyden S, Hames CG. The influence of increased dietary linoleate on essential hypertension in man. Acta Biol Med Ger. 1978;37(5-6):879-83. PMID 742306
- [Background] Comberg HU, Stern B: Blutdrucksenkung Bei Linolsaurereicher Diat-Zwei Pilotstudien. Aktuelle Ernahrungsmedizin in Klinik Und Praxis. Ban 3, Heft 5, Oct, 1978
- [Background] Graham TW, Kaplan BH, Cornoni-Huntley JC, James SA, Becker C, Hames CG, Heyden S. Frequency of church attendance and blood pressure elevation. J Behav Med. 1978 Mar;1(1):37-43. doi: 10.1007/BF00846585. PMID 556112
- [Background] Goust JM, Chenais F, Carnes JE, Hames CG, Fudenberg HH, Hogan EL. Abnormal T cell subpopulations and circulating immune complexes in the Guillain-Barre syndrome and multiple sclerosis. Neurology. 1978 May;28(5):421-5. doi: 10.1212/wnl.28.5.421. PMID 306075
- [Background] Farmer PK, Olewine DA, Comer DW, Edwards M, Coleman TM, Thomas G, Hames CG: Effect of Submaximal Exercise on Recovery Frontalis Muscle Tension and Occipital Alpha Wave Production in College-Aged Males. ASB Bulletin, 25:(No. 2), 87, Apr 1978
- [Background] Manegold Ch, Patzsche U: Serumkalium Bei 198 MIT Benzothiadiazin (Chlorthalidon) Behandelten Essentiellen Hypertonikern Wahrend Vier Jahren. Herz Keizlaug, 10, Nr. 12 (1978)
- [Background] Fleischman AI, Comberg HU, Hames CG. Platelet function and hypertension in humans. J Med Soc N J. 1979 Jan;76(1):17-20. No abstract available. PMID 284145
- [Background] Heyden S, Heiss G, Manegold C, Tyroler HA, Hames CG, Bartel AG, Cooper G. The combined effect of smoking and coffee drinking on LDL and HDL cholesterol. Circulation. 1979 Jul;60(1):22-5. doi: 10.1161/01.cir.60.1.22. PMID 221133
- [Background] Elston RC, Namboodiri KK, Hames CG. Segregation and linkage analyses of dopamine-beta-hydroxylase activity. Hum Hered. 1979;29(5):284-92. doi: 10.1159/000153059. PMID 489028
- [Background] Hames CG, Sauer HI. Cardiovascular disease death rates for counties in Georgia. J Med Assoc Ga. 1979 Nov;68(11):999-1001. No abstract available. PMID 501240
- [Background] Heyden S, Tyroler HA, Heiss G, Hames CG, Bartel A: Coffee Ingestion and Total Mortality Rates. Obesity Ger Med, 8:4, July-Aug, 1979
- [Background] Heyden S, Heyden F, Heiss G, Hames CG. Smoking and coffee consumption in three groups: cancer deaths, cardiovascular deaths and living controls. A prospective study in Evans County, Georgia. J Chronic Dis. 1979;32(9-10):673-7. doi: 10.1016/0021-9681(79)90098-5. No abstract available. PMID 489708
- [Background] Patzschke U, Manegold C. [Electrocardiographic signs of hypokalemia under antihypertensive treatment (author's transl)]. Schweiz Rundsch Med Prax. 1979 Jul 10;68(28):908-15. No abstract available. German. PMID 514983
- [Background] Patzschke U, Manegold Ch: Essentiele Hypertonie: Gestaltwandel Unter Antihypertensiver Behandlung. Diagnostik 12:167-169, 1979
- [Background] Manegold C, Patzschke U. [Regression of left ventricular hypertophy in the ECG during antihypertensive treatment: preliminary observations (author's transl)]. Dtsch Med Wochenschr. 1979 Jun 8;104(23):846-8. doi: 10.1055/s-0028-1104000. German. PMID 156115
- [Background] Patzschke U, Manegold C, Wolff G. [Reduction of hypertensive changes in the electrocardiogram during antihypertensive treatment]. MMW Munch Med Wochenschr. 1979 Jun 8;121(23):795-7. No abstract available. German. PMID 111073
- [Background] Grim CE, Luft FC, Miller JZ, Meneely GR, Battarbee HD, Hames CG, Dahl LK. Racial differences in blood pressure in Evans County, Georgia: relationship to sodium and potassium intake and plasma renin activity. J Chronic Dis. 1980;33(2):87-94. doi: 10.1016/0021-9681(80)90032-6. No abstract available. PMID 6986391
- [Background] Heyman A, Wilkinson WE, Heyden S, Helms MJ, Bartel AG, Karp HR, Tyroler HA, Hames CG. Risk of stroke in asymptomatic persons with cervical arterial bruits: a population study in Evans County, Georgia. N Engl J Med. 1980 Apr 10;302(15):838-41. doi: 10.1056/NEJM198004103021504. PMID 7360161
- [Background] Cutter G, Heyden S, Kasteler J, Kraus JF, Lee ES, Shipley T, Stromer M. Mortality surveillance in collaborative trials. Am J Public Health. 1980 Apr;70(4):394-400. doi: 10.2105/ajph.70.4.394. PMID 7361958
- [Background] Heyden S, Heiss G, Bartel AG, Hames CG. Sex differences in coronary mortality among diabetics in Evans County, Georgia. J Chronic Dis. 1980;33(5):265-73. doi: 10.1016/0021-9681(80)90021-1. No abstract available. PMID 7372764
- [Background] Dischinger P, Tyroler HA, McDonagh R Jr, Hames CG. Blood fibrinolytic activity, social class and habitual physical activity--I. A study of black and white men in Evans County, Georgia. J Chronic Dis. 1980;33(5):283-90. doi: 10.1016/0021-9681(80)90023-5. No abstract available. PMID 6445372
- [Background] Heyden S, Hames CG. Dietary effects on blood pressure. Nutr Metab. 1980;24 Suppl 1:50-64. doi: 10.1159/000176371. PMID 7454138
- [Background] Heyden S, Hames CG, Talton I. Potassium-rich foods - do they do the hypertensive patient any good? J Med Assoc Ga. 1980 May;69(5):395-7. No abstract available. PMID 7373178
- [Background] Heyden S, Heiss G, Hames CG, Bartel AG. Fasting triglycerides as predictors of total and CHD mortality in Evans County, Georgia. J Chronic Dis. 1980;33(5):275-82. doi: 10.1016/0021-9681(80)90022-3. No abstract available. PMID 7372765
- [Background] Tyroler HA, Heiss G, Schonfeld G, Cooper G, Heyden S, Hames CG. Apolipoprotein A-I, A-II and C-II in black and white residents of Evans County. Circulation. 1980 Aug;62(2):249-54. doi: 10.1161/01.cir.62.2.249. PMID 7397966
- [Background] Deubner DC, Wilkinson WE, Helms MJ, Tyroler HA, Hames CG. Logistic model estimation of death attributable to risk factors for cardiovascular disease in Evans County, Georgia. Am J Epidemiol. 1980 Jul;112(1):135-43. doi: 10.1093/oxfordjournals.aje.a112963. PMID 7395848
- [Background] Szczeklik A, Dischinger P, Kueppers F, Tyroler HA, Hames CG, Cassel JC, Creagan S. Blood fibrinolytic activity, social class and habitual physical activity--II. A study of black and white men in Southern Georgia. J Chronic Dis. 1980;33(5):291-9. doi: 10.1016/0021-9681(80)90024-7. No abstract available. PMID 6154717
- [Background] Heiss G, Tyroler HA, Gunnells JC, McGuffin WL, Hames CG. Dopamine-beta-hydroxylase in a biracial community: demographic, cardiovascular and familial factors. J Chronic Dis. 1980;33(5):301-10. doi: 10.1016/0021-9681(80)90025-9. No abstract available. PMID 7372766
- [Background] Kark JD, Smith AH, Hames CG. The relationship of serum cholesterol to the incidence of cancer in Evans County, Georgia. J Chronic Dis. 1980;33(5):311-32. doi: 10.1016/0021-9681(80)90026-0. No abstract available. PMID 7372767
- [Background] Tyroler HA: Editorial - John C. Cassel Memorial Symposium. J. Chronic Dis. 33:261, 1980
- [Background] Heyden S, Heiss G, Heyman A, Tyroler AH, Hames CG, Patzschke U, Manegold C. Cardiovascular mortality in transient ischemic attacks. Stroke. 1980 May-Jun;11(3):252-5. doi: 10.1161/01.str.11.3.252. PMID 7394861
- [Background] Pandey JP, Tung E, Mathur S, Namboodiri KK, Wang AC, Fudenberg HH, Blattner WA, Elston RC, Hames CG. Linkage relationship between variable and constant region allotypic determinants of human immunoglobulin heavy chains. Nature. 1980 Jul 24;286(5771):406-7. doi: 10.1038/286406a0. No abstract available. PMID 6772963
- [Background] Heyden S, Nelius SJ, Hames CG: Obesity, Salt Intake and Hypertension. J Cardiovasc Med. Nov, 1980
- [Background] Fogle TA, McKenzie WH. Cytogenetic study of a large black kindred: inversions, heteromorphisms, and segregation analysis. Hum Genet. 1980;55(3):345-52. doi: 10.1007/BF00290216. PMID 7203469
- [Background] Andrews JW, Hames CG, Metts JC Jr, Waters L, Davis JM, Carpenter R. Relationships between selenium and other parameters in drinking water and blood of subjects from high and low cardiovascular disease rate areas of Georgia. J Environ Pathol Toxicol. 1980 Sep;4(2-3):313-8. PMID 6970246
- [Background] Tyroler HA, Heiss G, Heyden S, Hames CG. Family follow-up study of serum cholesterol in Evans County, Georgia. J Chronic Dis. 1980;33(5):323-30. doi: 10.1016/0021-9681(80)90027-2. No abstract available. PMID 7372768
- [Background] Andrews J, Hames CG, Metts J, Davis J: Status of Selenium, Cadmium and Glutathione Peroxidase in Blood of Cardiovascular Diseased and Normal Subjects from Rural and Urban Area of the Cardiovascular Part of Southeastern United States. Trace Substances Environ Health, Vol 14, D.D. Hemphill, University of Missouri Press, 1980
- [Background] Fogle TA, Namboodiri KK, Elston RC, McKenzie WH, Hames CG. Linkage relationships of biochemical markers to Q- and C-band variants in a large black kindred. Hum Genet. 1980;55(3):353-6. doi: 10.1007/BF00290217. PMID 6937430
- [Background] Hames CG, Heyden S. Risk factors and hypertension. J Med Assoc Ga. 1981 May;70(5):337-8. No abstract available. PMID 7264465
- [Background] Patzschke U, Wolff Ch, Muhlbaier LH, Manegold Ch: Serumpipide Bei Essentiellen Hypertonikern Unter Chlortalidontherapie. Therapiewoche, 31:3405-3414, 1981
- [Background] Kark JD, Smith AH, Switzer BR, Hames CG. Serum vitamin A (retinol) and cancer incidence in Evans County, Georgia. J Natl Cancer Inst. 1981 Jan;66(1):7-16. PMID 6935468
- [Background] Kark JD, Smith AH, Switzer BR, Hames CG: Retinol, Carotene, and the Cancer Cholesterol Association. Lancet, June 20, 1981
- [Background] Kark JD, Smith AH, Hames CG. Serum retinol and the inverse relationship between serum cholesterol and cancer. Br Med J (Clin Res Ed). 1982 Jan 16;284(6310):152-4. doi: 10.1136/bmj.284.6310.152. PMID 6799076
- [Background] Kraus JF, Conley A, Hardy R, Sexton M, Sweezy Z. Relationship of demographic characteristics of interviewers to blood pressure measurements. J Community Health. 1982 Fall;8(1):3-12. doi: 10.1007/BF01324392. PMID 7186909
- [Background] Ockhuizen T, Pandey JP, Galbraith GM, Fudenberg HH, Hames CG. Autoantibodies and immunoglobulin allotypes in healthy North American Blacks of different age groups. Mech Ageing Dev. 1982 Jun;19(2):103-11. doi: 10.1016/0047-6374(82)90002-1. PMID 7109710
- [Background] Wing S, Aubert RE, Hansen JP, Hames CG, Slome C, Tyroler HA. Isolated systolic hypertension in Evans county--I. Prevalence and screening considerations. J Chronic Dis. 1982;35(9):735-42. doi: 10.1016/0021-9681(82)90097-2. PMID 7107806
- [Background] Hames CG: Opportunities for Research in Family Practice. Proceedings of the Georgia Rural Health Conference, Mercer University, Macon, Georgia, Oct. 21 and 22, 1982
- [Background] Parkerson GR Jr, Barr DM, Bass M, Bland CJ, Froom J, Geyman JP, Hames C, McWhinney I, Medalie JH, Moore AS, Perkoff G, Rosenblatt R, Seifert MH Jr, Spitzer W, Williams T, Wood M. Meeting the challenge of research in family medicine: report of The Study Group on Family Medicine Research. J Fam Pract. 1982 Jan;14(1):105-113. PMID 7054359
- [Background] Willett WC, Polk BF, Morris JS, Stampfer MJ, Pressel S, Rosner B, Taylor JO, Schneider K, Hames CG. Prediagnostic serum selenium and risk of cancer. Lancet. 1983 Jul 16;2(8342):130-4. doi: 10.1016/s0140-6736(83)90116-2. PMID 6134981
- [Background] Jenkins CD, Somervell PD, Hames CG. Does blood pressure usually rise with age? . . . Or with stress? J Human Stress. 1983 Sep;9(3):4-12. doi: 10.1080/0097840X.1983.9936124. PMID 6655235
- [Background] Halfon ST, Hames CG, Heyden S. Corneal arcus and coronary heart disease mortality. Br J Ophthalmol. 1984 Aug;68(8):603-4. doi: 10.1136/bjo.68.8.603. No abstract available. PMID 6743631
- [Background] Marazita ML, Elston RC, Namboodiri KK, Hames CG. Factors contributing to the variability in serum lipid levels and blood pressure in a large kindred. Am J Epidemiol. 1983 Dec;118(6):806-17. doi: 10.1093/oxfordjournals.aje.a113699. PMID 6650482
- [Background] Davis CE, Knowles M, Kark J, Heyden S, Hames CG, Tyroler HA: Serum Cholesterol Levels and Cancer Mortality: Evans County Twenty-Year Followup Study. Am Oil Chemist Soc, Chapt. 55, pp. 892-900, 1983
- [Background] Willett WC, Polk BF, Underwood BA, Stampfer MJ, Pressel S, Rosner B, Taylor JO, Schneider K, Hames CG. Relation of serum vitamins A and E and carotenoids to the risk of cancer. N Engl J Med. 1984 Feb 16;310(7):430-4. doi: 10.1056/NEJM198402163100705. PMID 6537988
- [Background] McAdam PA, Smith DK, Feldman EB, Hames C. Effect of age, sex, and race on selenium status of healthy residents of Augusta, Georgia. Biol Trace Elem Res. 1984 Feb;6(1):3-9. doi: 10.1007/BF02918316. PMID 24263742
- [Background] Wright JS, Dever GE. Mortality in rural Georgia. J Med Assoc Ga. 1984 May;73(5):283-7, 291. No abstract available. PMID 6736805
- [Background] Tyroler HA, Knowles MG, Wing SB, Logue EE, Davis CE, Heiss G, Heyden S, Hames CG. Ischemic heart disease risk factors and twenty-year mortality in middle-age Evans County black males. Am Heart J. 1984 Sep;108(3 Pt 2):738-46. doi: 10.1016/0002-8703(84)90667-7. PMID 6475743
- [Background] Heiss G, Schonfeld G, Johnson JL, Heyden S, Hames CG, Tyroler HA. Black-white differences in plasma levels of apolipoproteins: the Evans County Heart Study. Am Heart J. 1984 Sep;108(3 Pt 2):807-14. doi: 10.1016/0002-8703(84)90676-8. PMID 6433686
- [Background] Fudenberg HH, Whitten HD, Arnaud P, Khansari N, Tsang KY, Hames CG. Immune diagnosis of a subset of Alzheimer's disease with preliminary implications for immunotherapy. Biomed Pharmacother. 1984;38(6):290-7. PMID 6335404
- [Background] Hames CG: A study in Contrast - The Highest and Lowest Geographical Areas of Longevity in the U.S. Scien Jrnl of Ga Baptist Med Center, Vol. IV, No. 1, July, 1984
- [Background] Tyroler HA. Overview of risk factors for coronary heart disease in black populations. Am Heart J. 1984 Sep;108(3 Pt 2):658-60. doi: 10.1016/0002-8703(84)90651-3. PMID 6236685
- [Background] Peleg I, Heyden S, Knowles M, Hames CG. Serum retinol and risk of subsequent cancer: extension of the Evans County, Georgia, study. J Natl Cancer Inst. 1984 Dec;73(6):1455-8. PMID 6595454
- [Background] Tyroler HA, Hames CG: Hypertension and its Correlates in Relation to Twenty Year Mortality in Black Residents of Evans County, Ga. Saunders E, Hall WD, Shulman NB (Eds), in: Hypertension in Blacks; Epidemiology, Pathology, and Physiology and Treatment, Emory University School of Medicine, Chapter 3, 1985
- [Background] Baird DD, Tyroler HA, Heiss G, Chambless LE, Hames CG. Menopausal change in serum cholesterol. Black/white differences in Evans County, Georgia. Am J Epidemiol. 1985 Dec;122(6):982-93. doi: 10.1093/oxfordjournals.aje.a114202. PMID 3877458
- [Background] McAdam PA, Smith DK, Kuske TT, Teague RJ, Feldsman DS, Hames CG, Feldman EB: Selenium Status in Residents of Georgia, U.S.A. Nutr Res, Suppl 1, 144-146, 1985
- [Background] Curb JD, Borhani NO, Entwisle G, Tung B, Kass E, Schnaper H, Williams W, Berman R. Isolated systolic hypertension in 14 communities. Am J Epidemiol. 1985 Mar;121(3):362-70. doi: 10.1093/oxfordjournals.aje.a114007. PMID 4014125
- [Background] Curb JD, Borhani NO, Schnaper H, Kass E, Entwisle G, Williams W, Berman R. Detection and treatment of hypertension in older individuals. Am J Epidemiol. 1985 Mar;121(3):371-6. doi: 10.1093/oxfordjournals.aje.a114008. PMID 4014126
- [Background] Curb JD, Borhani NO, Blaszkowski TP, Zimbaldi N, Fotiu S, Williams W. Long-term surveillance for adverse effects of antihypertensive drugs. JAMA. 1985 Jun 14;253(22):3263-8. PMID 3999311
- [Background] Peleg I, Morris S, Hames CG. Is serum selenium a risk factor for cancer? Med Oncol Tumor Pharmacother. 1985;2(3):157-63. doi: 10.1007/BF02934543. PMID 4068802
- [Background] Heyden S, Borhani NO, Tyroler HA, Schneider KA, Langford HG, Hames CG, Hutchinson R, Oberman A. The relationship of weight change to changes in blood pressure, serum uric acid, cholesterol and glucose in the treatment of hypertension. J Chronic Dis. 1985;38(4):281-8. doi: 10.1016/0021-9681(85)90073-6. PMID 3889027
- [Background] Hudy SP, Caster WO, Hames CG: Changes in Food and Nutrient Intake Patterns Observed in Older Men and Women in Evans County, Ga. J Clin Exp Gerontology, 7 (2) 99-113, 1985
- [Background] Wing S, Manton KG, Stallard E, Hames CG, Tryoler HA. The black/white mortality crossover: investigation in a community-based study. J Gerontol. 1985 Jan;40(1):78-84. doi: 10.1093/geronj/40.1.78. PMID 3965564
- [Background] Johnson JL, Heineman EF, Heiss G, Hames CG, Tyroler HA. Cardiovascular disease risk factors and mortality among black women and white women aged 40-64 years in Evans County, Georgia. Am J Epidemiol. 1986 Feb;123(2):209-20. doi: 10.1093/oxfordjournals.aje.a114230. PMID 3946371
- [Background] Schoenbach VJ, Kaplan BH, Fredman L, Kleinbaum DG. Social ties and mortality in Evans County, Georgia. Am J Epidemiol. 1986 Apr;123(4):577-91. doi: 10.1093/oxfordjournals.aje.a114278. PMID 3953538
- [Background] Keil JE, Sutherland SE, Hames CG, Lackland DT, Gazes PC, Knapp RG, Tyroler HA. Coronary disease mortality and risk factors in black and white men. Results from the combined Charleston, SC, and Evans County, Georgia, heart studies. Arch Intern Med. 1995 Jul 24;155(14):1521-7. PMID 7605154
- [Background] Knapp RG, Schreiner PJ, Sutherland SE, Keil JE, Gilbert GE, Klein RL, Hames C, Tyroler HA. Serum lipoprotein(a) levels in elderly black and white men in the Charleston Heart Study. Clin Genet. 1993 Nov;44(5):225-31. doi: 10.1111/j.1399-0004.1993.tb03887.x. PMID 8313620
- [Background] White AD, Hames CG, Tyroler HA. Serum cholesterol and 20-year mortality in black and white men and women aged 65 and older in the Evans County Heart Study. Ann Epidemiol. 1992 Jan-Mar;2(1-2):85-91. doi: 10.1016/1047-2797(92)90041-n. PMID 1342269
- [Background] Hames CG, Rose K, Knowles M, Davis CE, Tyroler HA. Black-white comparisons of 20-year coronary heart disease mortality in the Evans County Heart Study. Cardiology. 1993;82(2-3):122-36. doi: 10.1159/000175863. PMID 8324775
- [Background] Arnett DK, Strogatz DS, Ephross SA, Hames CG, Tyroler HA. Greater incidence of electrocardiographic left ventricular hypertrophy in black men than in white men in Evans County, Georgia. Ethn Dis. 1992 Winter;2(1):10-7. PMID 1458211
- [Background] Hypertension Control in Black Women Would Have Major Health Impact: lntern Med News, July 15-31, 1986. (published interview).
- [Background] Check WA. Interdisciplinary efforts seek hypertension causes, prevention, therapy in blacks. JAMA. 1986 Jul 4;256(1):11-3, 17. doi: 10.1001/jama.256.1.11. No abstract available. PMID 3712703
- [Background] Olewine DA, Simpson MT, Jenkins CD, Ramsay FH, Zyzanski SJ, Thomas G, Hames CG: Catecholamines, Platelet Adhesiveness and the Coronary Prone. Psychiatric Spectator. VIII:No 5, April 1972
- [Background] Hames CG, Greenlund KJ. Ethnicity and cardiovascular disease: The Evans County heart study. Am J Med Sci. 1996 Mar;311(3):130-4. doi: 10.1097/00000441-199603000-00004. PMID 8615387